CLINICAL TRIAL: NCT07132424
Title: Determining the Relationship Between Foot Posture, Toe Flexor Strength, and Balance and Postural Control in Adolescents
Brief Title: Relationship Between Foot Posture, Toe Flexor Strength, and Balance in Adolescents
Status: Completed | Type: Observational
Sponsor: Istanbul Kültür University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Halenur Evrendilek, MSc PT, Istanbul Kültür University
Other Study IDs: 2025-06/06
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Adolescent; Foot Posture Index Score; Toe Flexor Strength; Flat Foot Acquired Bilateral (Pes Planus); Balance Assessment
Keywords: flat foot; toe muscle strength; balance; center of pressure
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Adolescents between 12-18 years old
  Interventions: Procedure: Assesment

INTERVENTIONS:
Procedure: Assesment — Foot posture, toe muscle strength and balance assesment

SUMMARY:
The foot plays a critical role in movement and postural control, with toe flexor strength linked to gait, performance, and stability. While these relationships are well studied in adults, evidence in adolescents is limited. Pes planovalgus may reduce push-off capacity and weaken postural responses through decreased toe muscle strength. This study aims to examine the relationship between foot posture, toe flexor strength, and balance, focusing on anterior-posterior center of pressure changes in adolescents.

DETAILED DESCRIPTION:
The foot, as the most distal part of the kinetic chain in contact with the ground, plays a key role in body movements and maneuvers. Toe flexor strength has been linked to gait speed, physical performance, and functional ability. Toe orientation and stability influence the center of pressure and surface adaptation, with the hallux being particularly important for postural control during weight shifts. While the relationship between toe strength and postural sway is established in adults, evidence in children and adolescents is limited. Pes planovalgus, characterized by a lowered medial longitudinal arch, can impair push-off mechanics and is associated with weaker toe muscles and poorer postural responses. However, the effect of foot posture and toe strength on anterior-posterior center of pressure changes-a marker of dynamic balance-remains unclear. This study aims to investigate the relationship between foot posture, toe flexor strength, balance, and postural control in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12-18 years, who have provided informed consent from both their guardian and themselves, will be included.

Exclusion Criteria:

* Individuals with acute lower extremity injury or pain
* Individuals with a history of lower extremity injury
* Individuals with leg length discrepancy
* Individuals diagnosed with scoliosis

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-08-20 (Actual); Primary Completion 2025-09-13 (Actual); Study Completion 2025-09-28 (Actual)

PRIMARY OUTCOMES:
Balance | Baseline
  Anterior-posterior (AP) center-of-pressure displacement and velocity will be calculated by collecting data with 2 force plates.
Foot Posture | Baseline
  Foot posture index - 6 will be used to determine foot posture of participants.
Toe muscle strength | Baseline
  Hallux and lesser toe flexor muscle strength will be assessed with a dynamometer while seated and pushing against it.
Navicular drop | Baseline
  Navicular drop will be used to assess foot posture.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Kultur University Motion Analysis Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided